CLINICAL TRIAL: NCT00893282
Title: A Randomized, Controlled, Prospective, Single Blind Clinical Evaluation of BackStop in Patients Undergoing Intraureteric Stone Lithotripsy.
Brief Title: Clinical Evaluation of BackStop in Patients Undergoing Intraureteric Stone Lithotripsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pluromed, Inc. (Industry)
Responsible Party: James Wilkie, Vice President, Operations, Pluromed, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BSTP-001
Record Dates: First submitted 2009-05-01; First posted 2009-05-05 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-05

CONDITIONS: Renal Calculi; Kidney Stones
Keywords: renal; calculi; kidney; stones
MeSH Terms: conditions — Kidney Calculi; Calculi

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- BackStop (Experimental): Intracorporeal lithotripsy with the use of an anti-retropulsion device.
  Interventions: Device: BackStop
- Control (Active Comparator): No anti-retropulsion device will be used during lithotripsy.
  Interventions: Device: Intracorporeal lithotripsy without the use of an anti-retropulsion device

INTERVENTIONS:
Device: BackStop — BackStop in a gel plug that potentially prevents retropulsion during intracorporeal lithotripsy.
  Arms: BackStop
Device: Intracorporeal lithotripsy without the use of an anti-retropulsion device
  Arms: Control

SUMMARY:
The purpose of this clinical study is to evaluate BackStop, a polymer-based device that is intended to be used during ureteroscopic lithotripsy to prevent retrograde stone migration. It is a water soluble polymer with reverse thermosensitive properties; the polymer exists as a liquid at low temperature (below 17 C) and rapidly transitions to a high viscosity gel at body temperature (i.e. in the ureter). BackStop is injected above the stones in the ureter and is intended to prevent retrograde migration of stones during ureteroscopic lithotripsy. Upon completion of the lithotripsy procedure, BackStop dissolves naturally or by irrigation.

The study hypothesis is that a greater proportion of patients will experience no retropulsion of a kidney stone when BackStop is used versus no anti-retropulsion device when undergoing intracorporeal lithotripsy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a solitary, radio-opaque ureteral stone in the proximal ureter.
* Clinical indication for treatment by ureteroscopic lithotripsy.
* Minimum 18 years old (or any institutional age limits for participation in clinical study).
* Patients must be willing and able to participate in any follow-up visits, as required.
* Patients must provide informed consent.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2008-02; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Ability of BackStop™ to minimize migration stone fragments in the proximal ureter will and reported as "yes" or "no". | intra-operative

SECONDARY OUTCOMES:
Extent of residual fragments remaining in ureter at the follow-up visit 2 to 4 weeks post-procedure. | one month
In the event that stone fragments migrate retrograde, there may be a need for the physician to employ additional procedures | one month

CONTACTS AND LOCATIONS:
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada